CLINICAL TRIAL: NCT05257135
Title: Development of a Prospective Clinico-biological Database in Cachexia in Patients With Colon Cancer
Brief Title: A Clinico-biological Database in Cachexia in Patients With Colon Cancer
Acronym: BCBCachexie
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2019-15-BCA
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological collection (Experimental): For all patients included in the study:
  * Blood samples collected at different times: at inclusion and during treatment every 6 months
  * In parallel to this biological collection, standardized clinical data will be entered into a database
  Interventions: Biological: Biological collection

INTERVENTIONS:
Biological: Biological collection — - Blood samples collected at different times: at inclusion and during treatment ( every 6 month)

SUMMARY:
Creation of a prospective clinico-biological database dedicated to cachexia and undernutrition in order to carry out future research projects, to improve our knowledge of colon cancer and cachexia and to optimize the therapeutic management of patients

DETAILED DESCRIPTION:
Patients with cancers, and in particular colorectal cancers, very often present profound nutritional and/or metabolic alterations, the most spectacular being cachexia. Cachexia is a morbid syndrome characterized by rapid involuntary weight loss mainly affecting the storage tissues of adipose tissue and skeletal muscle. This global metabolic syndrome is a major contributory factor and sometimes causative factor in the failure of treatments and the death of patients. Although a major public health problem, this disease is poorly understood and for which there are no reliable biomarkers and no universally accepted treatment protocol. It therefore appears essential to better understand this disease in order to improve the well-being and survival of patients. Being a disease with a strong metabolic component, the integration of nutritional approaches is essential. Many advances have been made in recent years in the field of clinical nutrition, particularly in cancer cachexia. Clinical nutrition is a new, transversal, booming specialty.

Recent publications suggests that cancer patients, overweight or obese, may present muscle depletion, an independent predictor of overall survival. Recent results suggest that muscle atrophy is associated with more severe toxicity of anti-cancer treatments such as fluoropyrimidines, anthracyclines, combination chemotherapy, sunitinib and sorafenib. Muscle wasting is a predictive factor for therapeutic dose limitation: dose reduction, delay or definitive discontinuation of treatment. The majority of anti-cancer drugs have a limited therapeutic index. It is important to determine the factors that explain the individual variations in efficacy and toxicity, and the determination of body composition for each patient is therefore an important step in the nutritional evaluation process, and essential data for this data base.

The investigators therefore propose the development of a prospective clinico-biological database for cachexia in patients with colon cancer, can be used for research projects aimed at developing tailored patient management strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old,
2. Patient treated at the Montpellier Regional Cancer Institute for colon cancer not eligible for surgery (of the primary tumor or associated metastases), whether undergoing treatment or not,
3. Patient requiring treatment for colon cancer (chemotherapy, targeted therapy, etc.),
4. Patient having accepted the constraints of the research and the blood samples planned for the research
5. Patient affiliated to Social Protection system
6. Informed consent form signed

Exclusion Criteria:

1. Patient requiring surgery (for treatment of colon cancer or metastasis)
2. Patient with exclusive peritoneal carcinomatosis
3. Patient requiring radiotherapy
4. Patient unable to understand or comply with study instructions or requirements for psychological, family, social or geographical reasons
5. Pregnant and/ or breastfeeding women
6. Patient cared for an emergency context

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Number of clinical risk factors for colorectal cancer | Until the study completion : 6 years
Number of biological risk factors for colorectal cancer | Until the study completion : 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Senesse, MD, Study Chair — Institut régional du cancer de Montpellier
Locations (1):
- Institut Régional du cancer de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chambrier C, Sztark F; Societe Francophone de nutrition clinique et metabolisme (SFNEP); Societe francaise d'anesthesie et reanimation (SFAR). French clinical guidelines on perioperative nutrition. Update of the 1994 consensus conference on perioperative artificial nutrition for elective surgery in adults. J Visc Surg. 2012 Oct;149(5):e325-36. doi: 10.1016/j.jviscsurg.2012.06.006. Epub 2012 Oct 26. PMID 23107793
- [Result] MacDonald AJ, Greig CA, Baracos V. The advantages and limitations of cross-sectional body composition analysis. Curr Opin Support Palliat Care. 2011 Dec;5(4):342-9. doi: 10.1097/SPC.0b013e32834c49eb. PMID 21986910
- [Result] Martin L, Birdsell L, Macdonald N, Reiman T, Clandinin MT, McCargar LJ, Murphy R, Ghosh S, Sawyer MB, Baracos VE. Cancer cachexia in the age of obesity: skeletal muscle depletion is a powerful prognostic factor, independent of body mass index. J Clin Oncol. 2013 Apr 20;31(12):1539-47. doi: 10.1200/JCO.2012.45.2722. Epub 2013 Mar 25. PMID 23530101
- [Result] Prado CM, Baracos VE, McCargar LJ, Mourtzakis M, Mulder KE, Reiman T, Butts CA, Scarfe AG, Sawyer MB. Body composition as an independent determinant of 5-fluorouracil-based chemotherapy toxicity. Clin Cancer Res. 2007 Jun 1;13(11):3264-8. doi: 10.1158/1078-0432.CCR-06-3067. PMID 17545532
- [Result] Prado CM, Sawyer MB, Ghosh S, Lieffers JR, Esfandiari N, Antoun S, Baracos VE. Central tenet of cancer cachexia therapy: do patients with advanced cancer have exploitable anabolic potential? Am J Clin Nutr. 2013 Oct;98(4):1012-9. doi: 10.3945/ajcn.113.060228. Epub 2013 Aug 21. PMID 23966429
- [Result] Antoun S, Baracos VE, Birdsell L, Escudier B, Sawyer MB. Low body mass index and sarcopenia associated with dose-limiting toxicity of sorafenib in patients with renal cell carcinoma. Ann Oncol. 2010 Aug;21(8):1594-1598. doi: 10.1093/annonc/mdp605. Epub 2010 Jan 20. PMID 20089558
- [Result] Baracos VE, Reiman T, Mourtzakis M, Gioulbasanis I, Antoun S. Body composition in patients with non-small cell lung cancer: a contemporary view of cancer cachexia with the use of computed tomography image analysis. Am J Clin Nutr. 2010 Apr;91(4):1133S-1137S. doi: 10.3945/ajcn.2010.28608C. Epub 2010 Feb 17. PMID 20164322